CLINICAL TRIAL: NCT01729143
Title: A Randomized, Cross-Over Trial to Evaluate the Acute Effects of Black Pepper on Energy Expenditure and Fat Oxidation in Humans
Brief Title: Impact of Black Pepper on Energy Expenditure and Substrate Utilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Appalachian State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 11-0468
Record Dates: First submitted 2012-11-13; First posted 2012-11-20 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2012-11

CONDITIONS: Obesity
Keywords: black pepper; metabolic chamber; respiratory chamber
MeSH Terms: conditions — Obesity | interventions — Energy Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Black pepper (Active Comparator): During the black pepper study day, subjects consumed 1.5g of black pepper (0.5g/meal) in 60.8g of vegetable juice. Black pepper was consumed was a meal on each occasion. 24-hour energy expenditure and substrate utilization will be measured.
  Interventions: Other: 24-hour energy expenditure and substrate utilization
- No pepper control (Placebo Comparator): During the no pepper control study day, subjects consumed an identical menu without black pepper. 60.8g of vegetable juice (vehicle) was consumed at each of the three study meals. 24-hour energy expenditure and substrate utilization will be measured.
  Interventions: Other: 24-hour energy expenditure and substrate utilization

INTERVENTIONS:
Other: 24-hour energy expenditure and substrate utilization — Subjects spent two x 24-hour periods inside the metabolic chamber at the UNC NRI (black pepper and no pepper control) each separated by one week. Subjects were requested to arrive at the study center each morning in a fasted state (at least 10 hours). During each study day, subjects remained sedentary. All meals were provided and were tailored to each subject's specific energy requirements. Study meals (with the exception of the 1.5g of black pepper) were identical between the black pepper and no pepper control study days.

SUMMARY:
As obesity rates worldwide continue to increase, there is a focus on identifying active food ingredients which increase metabolic rate which can be used as a dietary supplement in the treatment of overweight and obesity. Promising animal and cell studies have suggested a role for black pepper and an active component of black pepper, piperine, in energy expenditure. However, the effects of black pepper have not been determined in humans. The investigators hypothesis if that consumption of 1.5g black pepper (0.5g in each of three meals over one day) will result in an elevation in 24-h resting energy expenditure when contrasted to a control day (no black pepper, same diet intake).

ELIGIBILITY:
Inclusion Criteria:

* Woman
* Postmenopausal
* Aged 50-65 years
* BMI 25-35kg/m2
* Not taking blood pressure or anti-inflammatory medications or any other medications that may impact the results
* Thyroid hormone profile within the normal reference range
* No medical condition which may impact the results (e.g. diabetes)
* Accustomed to eating regular meals including breakfast

Exclusion Criteria:

* Smoker
* Heavy exerciser (defined as >150 minutes/week for more than 3 months)
* Abuses alcohol or drugs
* Vegetarian

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Energy expenditure and substrate oxidation | 24-hours
  A primary outcome of this study was the 24-hour energy expenditure (measured in the metabolic chamber at the UNC NRI) following black pepper and no pepper control.

SECONDARY OUTCOMES:
Gut peptides | 30 minutes after lunch
  Change in gut peptide secretion 30 minutes following a meal containing black pepper compared with no pepper control.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Swick, PhD, Principal Investigator — UNC Chapel Hill Nutrition Research Institute
Locations (1):
- UNC Chapel Hill Nutrition Research Institute, Kannapolis, North Carolina, United States

REFERENCES:
- [Derived] Swick AG, Orena S, O'Connor A. Irisin levels correlate with energy expenditure in a subgroup of humans with energy expenditure greater than predicted by fat free mass. Metabolism. 2013 Aug;62(8):1070-3. doi: 10.1016/j.metabol.2013.02.012. Epub 2013 Apr 8. PMID 23578923